CLINICAL TRIAL: NCT04554823
Title: Effects of a Physical Exercise and Health Education Program for Women With Breast Cancer Undergoing Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 328717
Record Dates: First submitted 2019-01-11; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Cancer, Breast
Keywords: Cancer; Physical Exercise; Health Education Program
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Verificar o efeito de um Programa de exercicios fisicos e de educacao em saude em mulheres com cancer de mama submetidas a quimioterapia sobre a taxa de conclusao da quimioterapia e sobre as toxicidades do tratamento.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Will attend lectures on health education.
  Interventions: Behavioral: Health Education; Behavioral: Physical Exercise
- Exercise Group (Experimental): Will be subjected to a supervised training program of combined exercises for 24 weeks, with a frequency of 3 times weekly and duration of 60 minutes, an unsupervised flexibility training program 2 times a week and Will attend lectures on health education.
  Interventions: Behavioral: Health Education; Behavioral: Physical Exercise

INTERVENTIONS:
Behavioral: Health Education — Will attend lectures on health education about Health and Physical Education, healthy eating, overcoming barriers, Back to routine, Physical Activity Options and Dealing with Stress and Depression
Behavioral: Physical Exercise — Supervised physical training program of combined exercises for 24 weeks, with frequency of 3 times weekly and duration of 60 minutes, an unsupervised flexibility training program 2 times a week.

SUMMARY:
The purpose of this study is to verify the effect of the intervention of a program of physical exercises and health education in women with breast cancer undergoing chemotherapy.

DETAILED DESCRIPTION:
According to the National Cancer Institute (INCA), the estimate for Brazil, 2016-2017 biennium, points to the occurrence of about 600,000 new cases of cancer, and breast cancer (58000) in women will be the most frequent. One study revealed that only 12% of women undergoing chemotherapy in CM who participated in a physical exercise program had to readjusted the dose of the medications, while 34% of those who received the conventional treatment needed to readjust the Treatment doses, with neuropathy being one of the most present adverse effects that influenced this adjustment. In this sense, the conduct to keep the patient at rest during the treatment seems to potentiate her side effects, and sedentarism is another factor detrimental to the patient's health. Objective: To verify the effect of the intervention of a program of physical exercises and health education in women with breast cancer undergoing chemotherapy. Methodology: A sample will consist of 136 (136) Women, over 18 years of age, sedentary, diagnosed with non-metastatic breast cancer and initiating the first cycle of chemotherapy. They will be divided into two groups, randomly and stratified: control group: (CG n = 68) and exercise group: (eg n = 68) that will undergo a supervised training program of combined exercises for 24 weeks, with a frequency of 3 times Weekly and duration of 60 minutes, an unsupervised flexibility training program 2 times a week and both groups (GC and EG) will attend lectures on health education, which are held monthly.

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years of age;
* with the first diagnosis of non-metastatic breast cancer;
* Sedentary for 6 months;
* who are in the initial cycle of chemotherapy;
* with the release of the responsible physician;
* availability to participate in the exercise program;
* signing of the free and clarified consent term.

Exclusion Criteria:

* women with clinical risk for physical exercise (e.g. severe anemia, ICC, CRI);
* Pregnant women;
* Osteoarticular problems that preclude the practice of physical exercise.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy completion rate | 6 months
  Effect of physical training on the rate of chemotherapy completion in the anthropometric profile, habitual food consumption, prevalence of comorbidities, cardiovascular, neurofunctional, bone and respiratory toxicity, myelosuppression, sarcopenia induced by chemotherapy, myalgia, nausea and vomiting symptoms.
Analysis of the level of Quality of Life | 6 months
  effect of physical training on the level of physical activity, perception of fatigue and pain, mood, sexual life, anxiety and depression and body image.
Physical aptitude | 6 months
  Effect of physical training during adjuvant and neoadjuvant chemotherapy on the levels of fragility, muscle strength, joint amplitude of the shoulder and cardiorespiratory capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Mayra Trevisani, Study Chair — External Researcher; Luana Queiroga, Study Chair — Employee
Locations (1):
- Hospital Municipal Vila Santa Catarina, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No